CLINICAL TRIAL: NCT06751550
Title: Change in Daily FeNO During Three Weeks of Inpatient Pulmonary Rehabilitation in Patients with Asthma
Brief Title: Changes in FeNO Value During Pulmonary Rehabilitation in Patients with Asthma
Acronym: Asthma FeNO
Status: Completed | Type: Observational
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Collaborators: Bosch Healthcare Solutions GmbH (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Andreas Rembert Koczulla, Professor, Schön Klinik Berchtesgadener Land
Other Study IDs: 168/20
Record Dates: First submitted 2024-12-20; First posted 2024-12-30 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Asthma Bronchiale; Asthmatic Patients; Asthmatics
Keywords: FeNO; Fractional Exhaled Nitric Oxide
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Asthmatic patients

SUMMARY:
This study investigates the use of fractional exhaled nitric oxide (FeNO) measurement to monitor non-pharmacological therapy during a three-week inpatient rehabilitation programme for asthma patients. It compares FeNO levels (measured three times a day) with clinical parameters and quality of life to analyse daily fluctuations and the acute effect of exercise training on FeNO levels. As FeNO is a non-invasive biomarker of airway inflammation, this study aims to expand its role in therapy monitoring and explore its application in a rehabilitation setting.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of bronchial asthma (all disease severities)
* Chronic Obstructive Pulmonary Disease (COPD) with an asthma component, where the asthma component plays a clinically relevant role
* written informed consent

Exclusion Criteria:

* Chronic Obstructive Pulmonary Disease (COPD) as the primary disease
* unability to perform FeNO measurement independently

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruitet at the pulmonary rehabilitation center at the Schön Klinik Berchtesgadener Land in Schönau am Königssee, Germany
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Fractional Exhaled Nitric Oxide (FeNO) at rest | From enrollment to the end of rehabilitation at 3 weeks. Daily measurements at 9AM; 1PM; 5PM
  Measurement of FeNo will be done with the Vivatmo Me device (by Bosch Health Care Solutions GmbH)
Fractional Exhaled Nitric Oxide (FeNO) before/after exercise | From enrollment to the end of rehabilitation at 3 weeks, FeNO measurements will be done before and after a bicycle endurance training
  Measurement of FeNo will be done with the Vivatmo Me device (by Bosch Health Care Solutions GmbH)

SECONDARY OUTCOMES:
Asthma control | On admission and discharge from the 3-week rehabilitation programme
  Assessed by Asthma Control Test (ACT)
Lung function | On admission and discharge from the 3-week rehabilitation programme
  Forced expiratory flow in 1 second, will be measured by Bodyplethysmography
Eosinophils | On admission and discharge from the 3-week rehabilitation programme
  Eosinophils will be collected by venous blood sample. Unit: total number of cells per ul blood and percentage
C-reactive protein | On admission and discharge from the 3-week rehabilitation programme
  C-reactive protein will be collected by venous blood sample. Unit: mg/liter
Immunoglobulin E (IgE) | On admission and discharge from the 3-week rehabilitation programme
  Immunoglobulin E will be collected by venous blood sample. Unit: ug/liter
6-minute walk test | On admission and discharge from the 3-week rehabilitation programme
  This test will be performed according to the described standard of the American Thoracic Society and the European Respiratory Society 2014

CONTACTS AND LOCATIONS:
Locations (1):
- Schön Klinik Berchtesgadener Land, Schönau am Königssee, Germany

IPD SHARING:
Plan to Share IPD: Yes
The data will be made available upon personal request.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be made available upon personal request.
Access Criteria: The data will be made available upon personal request submitting a proposal that describes planned analyses.